CLINICAL TRIAL: NCT05675800
Title: Psilocybin for the Treatment of Major Depressive Disorder
Brief Title: Psilocybin for Major Depressive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Resident who was tasked with coordinating this study is no longer able to do so.
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ginger E Nicol, Associate Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209153; R25MH112473 (NIH)
Record Dates: First submitted 2022-11-22; First posted 2023-01-09 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin Active Dose Treatment A (Experimental): Psilocybin
  Interventions: Drug: Psilocybin
- Psilocybin Active Dose Treatment B (Experimental): Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin administered with psychological support

SUMMARY:
The goal of this study is to assess the effectiveness of psilocybin for the treatment of Major Depressive Disorder and potential therapeutic mechanisms. Enrolled participants will receive a single active dose of psilocybin, or a dose considered high enough to treat depression, administered orally with accompanying psychological support.

ELIGIBILITY:
Inclusion Criteria:

* Currently meeting DSM-V Criteria for a Major Depressive Episode of at least mild-moderate severity
* Aged 18-85
* Ability and willingness to attend study visits and complete study assessments

Exclusion Criteria:

* Presence of medical conditions at screening that may affect the safe administration of psilocybin (including, but not limited to: AST/ALT > 150, QTc > 450ms, MELD > 9)
* Depression deemed secondary to a severe medical condition
* Recent use of any classical psychedelic drug or MDMA
* Recent use of any interventional psychiatric treatment (including: ECT, ketamine, esketamine, TMS)
* Intention to begin any new treatment for depression prior to primary outcome determination
* Use of any excluded medication
* Active substance use disorder
* Presence of any psychiatric condition that may interfere with the safe administration of psilocybin
* Active suicidal ideation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
MADRS (Montgomery-Asberg Depression Rating Scale) Change from Baseline | 3 weeks post-treatment
  Depression severity rating scale, range 0-60 with higher scores indicating more severe symptoms
Adverse Events | Up to 12 weeks post-treatment
  Rates of adverse events related to treatment, as determined by multiple data collection mechanisms
Study Retention and Completion | Throughout study participation (12-17 weeks)
  Rates of successful attendance of study visits and completion of study

SECONDARY OUTCOMES:
MADRS (Montgomery-Asberg Depression Rating Scale) Change from Baseline | 12 weeks post-treatment
  Depression severity rating scale, range 0-60 with higher scores indicating more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and analysis plan will be publicly available on publication of the research. Individual researchers can request individual participant data collected during the trial, after deidentification, for specifically outlined research-related purposes upon publication.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication, indefinitely
Access Criteria: Investigators with a research plan that is reviewed and approved by the P.I.